CLINICAL TRIAL: NCT02087943
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Efficacy and Safety Study of Apremilast (CC-10004) in Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Study of Apremilast in Subjects With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CC-10004-AD-001
Record Dates: First submitted 2014-03-13; First posted 2014-03-14 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2017-04

CONDITIONS: Dermatitis, Atopic Dermatitis
Keywords: Atopic Dermatitis; Atopic Eczema
MeSH Terms: conditions — Dermatitis, Atopic | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Apremilast 40 mg (Experimental): Apremilast 40 mg administered orally twice daily (BID) for 12 weeks (following dose titration) during the placebo controlled phase followed by 40 mg Apremilast tablets orally administered BID for an additional 12 weeks in the active treatment phase
  Interventions: Drug: Apremilast
- Apremilast 30 mg (Experimental): Apremilast 30 mg administered orally BID for 12 weeks (following dose titration) during the placebo controlled phase followed by 30 mg Apremilast tablets orally administered BID for an additional 12 weeks in the active treatment phase
  Interventions: Drug: Apremilast
- Placebo + Apremilast 40 mg (Experimental): Placebo administered orally BID for 12 weeks, during the placebo controlled phase followed by 40 mg Apremilast tablets orally BID for an additional 12 weeks in the active treatment phase
  Interventions: Drug: Apremilast; Drug: Placebo
- Placebo + Apremilast 30 mg (Experimental): Placebo administered orally BID for 12 weeks, during the placebo controlled phase followed by 30 mg Apremilast tablets orally BID for an additional 12 weeks in the active treatment phase
  Interventions: Drug: Apremilast; Drug: Placebo
- Placebo (Placebo Comparator): Oral Placebo tablets administered twice daily (BID) for 12 weeks during the placebo-controlled phase.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Orally twice a day (BID)
  Other Names: CC-10004; Otezla
  Arms: Apremilast 40 mg; Placebo + Apremilast 40 mg
Drug: Apremilast — Orally twice a day (BID)
  Other Names: CC-10004; Otezla
  Arms: Apremilast 30 mg; Placebo + Apremilast 30 mg
Drug: Placebo — Orally twice a day (BID)
  Arms: Placebo + Apremilast 40 mg
Drug: Placebo — Orally twice a day (BID)
  Arms: Placebo; Placebo + Apremilast 30 mg

SUMMARY:
A study to evaluate the efficacy and safety of apremilast (CC-10004) in subjects with moderate to severe atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged ≥ 18 years (≥ 20 for Japanese subjects) at the time of consent.
2. Have a diagnosis of atopic dermatitis for ≥ 12 months.
3. Have moderate to severe atopic dermatitis which is considered inappropriate for topical therapy or which cannot be adequately controlled by topical therapy.
4. Meet the laboratory criteria as defined per protocol
5. Females of Childbearing Potential (FCBP) must have a negative pregnancy test at Screening and Baseline. Sexually active FCBP must use one of the approved contraceptive options required per protocol while on and for at least 28 days after the last dose of study medication
6. Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception while on and for at least 28 days after the last dose of study medication.

Exclusion Criteria:

1. Active tuberculosis (TB) or a history of inadequately treated tuberculosis.
2. Positive for hepatitis B surface antigen or hepatitis C antibody
3. Pregnant or breast feeding
4. History of allergy to any component of the study medication.
5. Active skin infection requiring systemic antimicrobials at Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- United States (15):
  - Arizona Research Center, Phoenix, Arizona
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Dermatology Research Associates, Los Angeles, California
  - Renstar Medical Research, Ocala, Florida
  - Emory Clinic, Atlanta, Georgia
  - Advanced Medical Research, Atlanta, Georgia
  - Northwestern University Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Dermatology Specialists, PSC, Louisville, Kentucky
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Department of Dermatology, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - PMG Research of Winston-Salem LLC, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Virginia Clinical Research Inc, Norfolk, Virginia
- Canada (6):
  - Chih-Ho Hong Medical, Inc., Surrey, British Columbia
  - Eastern Canada Cutaneous Research Associates Ltd, Halifax, Nova Scotia
  - Ultranova Skincare, Barrie, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm Research, Montreal, Quebec
  - Centre Dermatologique du Quebec Metropolitain, Ste-Foy, Quebec
- Japan (10):
  - Kokubu Abashiri Dermatology Clinic, Abashiri-shi, Hokkaido
  - Asanuma Dermatology Clinic, Chitose-shi, Hokkaido
  - Fukuoka University Hospital Dermatology, Fukuoka-shi, Fukuoka
  - Hatamoto Dermatology Clinic, Fukuoka-shi, Fukuoka
  - Tashiro Clinic, Iizuka-shi, Fukuoka
  - Kokubu Dermatology, Kitami-shi, Hokkaido
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Sapporo Skin Clinic, Sapporo-shi, Hokkaido
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Simpson EL, Imafuku S, Poulin Y, Ungar B, Zhou L, Malik K, Wen HC, Xu H, Estrada YD, Peng X, Chen M, Shah N, Suarez-Farinas M, Pavel AB, Nograles K, Guttman-Yassky E. A Phase 2 Randomized Trial of Apremilast in Patients with Atopic Dermatitis. J Invest Dermatol. 2019 May;139(5):1063-1072. doi: 10.1016/j.jid.2018.10.043. Epub 2018 Dec 5. PMID 30528828

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment assignment was stratified by geographic region and within each region, by the Eczema Area and Severity Index (EASI) score (≤ 20 or > 20). Six participants were excluded from analysis due to unsigned case books; a total of 185 participants were included in the final analyses.
Groups:
- Placebo: Participants initially randomized to identically matching placebo (PBO) tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-12)
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled phase and continued to receive 30 mg apremilast tablets twice daily (BID) for up to Week 24 in the active treatment phase
- Apremilast 40 mg: Participants initially randomized to receive 40 mg apremilast tablets twice daily in the 12-week placebo-controlled phase and continued to receive 40 mg apremilast tablets twice daily (BID) for up to Week 24 in the active treatment phase.
- Placebo/Apremilast 30 mg: Participants initially randomized to identically matching placebo tablets twice daily and were re-randomized at Week 12 to 30 mg apremilast for 12 weeks, up to week 24.
- Placebo/Apremilast 40 mg: Participants initially randomized to identically matching placebo tablets twice daily and were re-randomized at Week 12 to 40 mg apremilast for 12 weeks, up to week 24.
Period: Placebo-Controlled Phase Week 0-12
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Placebo/Apremilast 30 mg | Placebo/Apremilast 40 mg
Started | 64 | 58 | 63 | 0 | 0
Safety Population | 64 (Includes all participants who received at least one dose of study drug.) | 58 (Includes all participants who received at least one dose of study drug.) | 63 (Includes all participants who received at least one dose of study drug.) | 0 | 0
Completed | 50 (3 participants who completed week 12 did not enter the active treatment phase.) | 46 | 50 (1 participant who completed week 12 did not enter the active treatment phase.) | 0 | 0
Not Completed | 14 | 12 | 13 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 6 | 0 | 0
Not completed — Lack of Efficacy | 8 | 7 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Period: Active Treatment Phase Week 12-24
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Placebo/Apremilast 30 mg | Placebo/Apremilast 40 mg
Started | 0 | 46 | 49 | 24 | 23
Completed | 0 | 42 | 44 | 22 | 21
Not Completed | 0 | 4 | 5 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Other-Unspecified | 0 | 0 | 1 | 1 | 0
Period: Observational Follow-up Phase Week 24-30
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Placebo/Apremilast 30 mg | Placebo/Apremilast 40 mg
Started | 0 | 46 | 48 | 24 | 23
Completed | 0 | 46 | 45 | 23 | 22
Not Completed | 0 | 0 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) includes all participants who were randomized as specified in the protocol and received at least one dose of Investigational product (IP)
Groups:
- Placebo: Participants initially randomized to identically matching placebo (PBO) tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-16)
- Apremilast 30 mg: Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled phase.
- Apremilast 40 mg: Participants initially randomized to receive 40 mg apremilast tablets twice daily in the 12-week placebo-controlled phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg | Total
Number analyzed (Participants) | 64 | 58 | 63 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (14.71) | 39.2 (15.80) | 38.3 (14.74) | 38.4 (15.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 27 | 32 | 98
  Male | 25 | 31 | 31 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in the Eczema Area and Severity Index (EASI) Score at Week 12.
Description: EASI is a validated composite scoring system integrating the proportion of the body region (area) involved and the intensity of key signs of atopic dermatitis (AD). A representative lesion is selected for each of the four body regions for assessing the intensity of each of the four signs (erythema, induration /papulation, excoriation, and lichenification). Symptoms (eg, pruritus) and secondary signs (eg, xerosis, scaling) are excluded from the assessment. The total EASI score ranges from 0 to 72. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Time Frame: Baseline to Week 12
Population: All participants who were randomized as specified per protocol and who received at least one dose of IP with a baseline and at least 1 post baseline value at or before week 12; A missing value at Week 12 was imputed by last observation carried forward (LOCF), including the value obtained at the Early Termination Visit prior to Week 12.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 62 | 58 | 63
percent change | -10.98 (6.873) | -25.99 (7.106) | -31.57 (6.820)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.1308, ANCOVA — Based on an analysis of covariance model with the percentage change from baseline as the response variable and the treatment group and Baseline EASI score stratification (≤ 20, > 20) as factors; LS Mean Difference = -15.01, 95% CI 2-sided [-34.52 to 4.50]
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority or Other; p = 0.0347, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -20.60, 95% CI 2-sided [-39.70 to -1.50]

2. Secondary Outcome: Percentage of Participants Who Achieved a Score of 0 (Cleared) or 1 (Almost Cleared) and at Least a 2-point Reduction From Baseline in a Static Physician's Global Assessment of Acute Signs (sPGA-A) at Week 12.
Description: The sPGA-A is intended to assess the global severities (ie, a "visual average" integrating all areas of AD) of key acute clinical signs of AD, including erythema, induration/papulation, oozing/crusting (lichenification excluded) based on a 5-point scale of cleared (0), almost cleared (1), mild (2), moderate (3) and severe (4).
Time Frame: Baseline to Week 12
Population: ITT includes all participants who were randomized as specified per protocol and received at least one dose of IP. LOCF for missing data handling.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 64 | 58 | 63
percentage of participants | 6.3 | 3.4 | 14.3
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.4938, Cochran-Mantel-Haenszel — Adjusted treatment differences in proportions using the weighted average of the treatment differences across the stratum of baseline EASI score stratification (≤ 20, > 20) with, Cochran-Mantel-Haenszel (CMH) weights; Adjusted Difference in Proportion = -2.7, 95% CI 2-sided [-10.2 to 4.8] — 2-sided 95% Confidence Intervals (CI) is based on a normal approximation to the weighted average
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority or Other; p = 0.1368, Cochran-Mantel-Haenszel — Adjusted treatment differences in proportions using the weighted average of the treatment differences across the stratum of baseline EASI score stratification (≤ 20, > 20) with, CMH weights; Adjusted Difference in Proportion = 8.0, 95% CI 2-sided [-2.3 to 18.2] — 2-sided 95% Confidence Intervals (CI) is based on a normal approximation to the weighted average

3. Secondary Outcome: Percentage of Participants Who Achieved at Least a 50% Reduction From Baseline in the EASI Score (EASI 50) at Week 12
Description: The EASI 50 reduction (defined as ≥ 50% reduction from baseline in EASI score) was selected to serve as the key responder endpoint. A ≥ 50% improvement is clinically meaningful for this population.
Time Frame: Baseline to Week 12
Population: ITT includes all participants who were randomized as specified in the protocol and received at least one dose of IP. LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 64 | 58 | 63
percentage of participants | 32.8 | 31.0 | 42.9
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.8589, Cochran-Mantel-Haenszel; Adjusted Difference in Proportion = -1.5, 95% CI 2-sided [-18.0 to 14.9] — Adjusted differences in proportions was the weighted average of the treatment differences across the stratum of baseline EASI score stratification (≤ 20, > 20) with the CMH weights
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority or Other; p = 0.2476, Cochran-Mantel-Haenszel; Adjusted Difference in Proportion = 9.9, 95% CI 2-sided [-6.7 to 26.6] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: The Percentage Change From Baseline in the Average Weekly Pruritus Numerical Rating Scale (NRS) Score at Week 4
Description: The participant completed a daily diary recording the average intensity of pruritus they experienced during the preceding 24 hrs. The intensity of pruritus was assessed using a validated 11-point NRS, ranging from 0 ("no pruritus") to 10 ("the worst pruritus imaginable"). It should be noted that this NRS is distinct from the pruritus, Visual Analogue Scale (VAS) in the Modified SCORAD Index with respect to recall period (three days for the VAS). The weekly NRS score was calculated as the average of the NRS scores over 7 days within the specified week. A higher score indicated worse disease status, and a negative change from baseline indicated improvement.
Time Frame: Baseline to Week 4
Population: All participants who were randomized as specified in the protocol and who received at least one dose of IP with a baseline and at least 1 postbaseline value at or before Week 4 were included. LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 63 | 58 | 59
percent change | -4.83 (5.657) | -10.00 (5.911) | -9.00 (5.850)
Statistical Analysis 1: Comparison: Placebo vs Apremilast 30 mg; Test type: Superiority or Other; p = 0.5286, ANCOVA; LS Mean Difference = -5.17, 95% CI 2-sided [-21.34 to 10.99] — Based on an analysis of covariance model with the percentage change from baseline as the response variable, treatment group and baseline EASI stratification (≤ 20, > 20) as factors, and the baseline average weekly pruritus NRS score as a covariate
Statistical Analysis 2: Comparison: Placebo vs Apremilast 40 mg; Test type: Superiority or Other; p = 0.6092, ANCOVA; LS Mean Difference = -4.17, 95% CI 2-sided [-20.22 to 11.88] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During the Placebo Controlled Period
Description: A TEAE is an adverse event with a start date on or after the date of the first dose of IP and no later than 28 days after the last dose of IP for participants who discontinued early. An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre existing condition) should be considered an AE. A serious AE is any which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect; constitutes an important medical event.
Time Frame: Baseline to Week 12
Population: Safety population includes all participants who received at least one dose of IP.
Measure: Number; unit: participants
Arm/Group | Placebo | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 64 | 58 | 63
participants
  TEAE | 30 | 36 | 44
  Drug-related TEAE | 8 | 26 | 27
  Severe TEAE | 0 | 0 | 1
  Serious TEAE (SAE) | 0 | 1 | 2
  Drug-related SAE | 0 | 0 | 1
  TEAE Leading to Drug Interruption | 3 | 0 | 4
  TEAE Leading to Drug Withdrawal | 1 | 2 | 6
  Death | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With TEAEs During the Apremilast Exposure Period
Description: A TEAE is an adverse event with a start date on or after the date of the first dose of investigational product (IP) and no later than 28 days after the last dose of IP. An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre existing condition) should be considered an AE. A serious AE is any which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect; constitutes an important medical event.
Time Frame: Baseline to Week 24; median duration of apremilast 30 mg was 23.3 weeks and 22.4 weeks for apremilast 40 mg
Population: Safety population includes all participants who received at least one dose of IP. These were Apremilast participants as treated.
Measure: Number; unit: participants
Groups:
- Apremilast 30 mg: Participants initially randomized to 30 mg apremilast tablets twice daily in the 12-week placebo-controlled phase and continued receiving 30 mg apremilast tablets twice daily (BID) up to Week 24 in the active treatment, and for participants who were initially randomized to placebo and at week 12 subsequently randomized to 30 mg apremilast tablets twice daily in the active treatment phase.
- Apremilast 40 mg: Participants initially randomized to 40 mg apremilast tablets twice daily in the 12-week placebo-controlled phase and continued receiving 40 mg apremilast tablets twice daily (BID) up to Week 24 in the active treatment phase, and for participants who were initially randomized to placebo and at week 12 subsequently randomized to 40 mg apremilast tablets twice daily in the active treatment phase.
Arm/Group | Apremilast 30 mg | Apremilast 40 mg
Number analyzed (Participants) | 82 | 86
participants
  TEAE | 49 | 61
  Drug-related TEAE | 29 | 38
  Severe TEAE | 1 | 1
  Serious TEAE (SAE) | 2 | 3
  Drug-related SAE | 0 | 2
  TEAE Leading to Drug Interruption | 0 | 8
  TEAE Leading to Drug Withdrawal | 3 | 9
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events are reported for the 12-week placebo-controlled phase and up to 24 weeks for all participants who received apremilast at any time during the study. All TEAEs were recorded by the investigator from the time the participant received the first dose of study drug to no later than 28 days after the last dose of study drug.
Groups:
- Placebo (Weeks 0-12): Participants initially randomized to identically matching PBO tablets twice daily BID during the Placebo-controlled Phase (Weeks 0-12)
- Apremilast 30 mg (Weeks 0-12): Participants initially randomized to receive 30 mg apremilast tablets twice daily in the 12-week placebo-controlled phase.
- Apremilast 40 mg (Weeks 0-12): Participants initially randomized to receive 40 mg apremilast tablets twice daily in the 12-week placebo-controlled phase.
- Apremilast 30 mg (Apremilast Exposure Period) 0-24: Participants who received 30 mg PO BID apremilast, regardless of when the apremilast exposure started (at Week 0 or at Week 12 up until Week 24.
- Apremilast 40 mg (Apremilast Exposure Period) 0-24: Participants who received 40 mg PO BID apremilast, regardless of when the apremilast exposure started (at Week 0 or at Week 12 up until Week 24.
Arm/Group | Placebo (Weeks 0-12) | Apremilast 30 mg (Weeks 0-12) | Apremilast 40 mg (Weeks 0-12) | Apremilast 30 mg (Apremilast Exposure Period) 0-24 | Apremilast 40 mg (Apremilast Exposure Period) 0-24
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/58 | 2/63 | 2/82 | 3/86
Other Adverse Events (participants affected / at risk) | 14/64 | 22/58 | 30/63 | 30/82 | 45/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-12) (N=64) | Apremilast 30 mg (Weeks 0-12) (N=58) | Apremilast 40 mg (Weeks 0-12) (N=63) | Apremilast 30 mg (Apremilast Exposure Period) 0-24 (N=82) | Apremilast 40 mg (Apremilast Exposure Period) 0-24 (N=86)
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Weeks 0-12) (N=64) | Apremilast 30 mg (Weeks 0-12) (N=58) | Apremilast 40 mg (Weeks 0-12) (N=63) | Apremilast 30 mg (Apremilast Exposure Period) 0-24 (N=82) | Apremilast 40 mg (Apremilast Exposure Period) 0-24 (N=86)
Nasopharyngitis (Infections and infestations) | 1 | 6 | 6 | 8 | 14
Upper respiratory tract infection (Infections and infestations) | 8 | 2 | 3 | 8 | 6
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 0 | 5
Headache (Nervous system disorders) | 5 | 4 | 8 | 7 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 10 | 15 | 11 | 21
Nausea (Gastrointestinal disorders) | 1 | 9 | 7 | 10 | 14
Abdominal discomfort (Gastrointestinal disorders) | 0 | 3 | 2 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 1 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 12 months since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 days. Investigator must delete confidential information before submission or defer publication to permit patent applications.